CLINICAL TRIAL: NCT04434937
Title: A Phase 2, Multicenter, Open-Label Study of Parsaclisib, a PI3Kδ Inhibitor, in Japanese Participants With Relapsed or Refractory Follicular Lymphoma (CITADEL-213)
Brief Title: Open-Label Study of Parsaclisib, in Japanese Participants With Relapsed or Refractory Follicular Lymphoma (CITADEL-213)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Biosciences Japan GK (Industry)
Responsible Party: Sponsor
Organization: Incyte Corporation (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCB 50465-213
Record Dates: First submitted 2020-06-15; First posted 2020-06-17 (Actual); Results first posted 2024-01-03 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-08

CONDITIONS: Lymphoma
Keywords: Follicular Lymphoma; Parsaclisib; PI3Kδ Inhibitor
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular | interventions — parsaclisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- parsaclisib (Experimental): parsaclisib will be taken orally QD with water without regard to food except on mornings of PK clinic visits
  Interventions: Drug: parsaclisib

INTERVENTIONS:
Drug: parsaclisib — parsaclisib will be taken orally QD with water without regard to food except on mornings of PK clinic visits
  Other Names: INCB050465

SUMMARY:
The purpose of this study is to assess the efficacy and safety of parsaclisib in Japanese participants with relapsed or refractory follicular lymphoma

ELIGIBILITY:
Inclusion Criteria:

* Male or female Japanese participant who must be ≥ 18 years of age
* Ability to comprehend and willingness to sign a written ICF and comply with all study visits and procedures
* Histologically confirmed, relapsed or refractory, FL Grade 1, 2, and 3a
* Ineligible for HSCT
* Must have been treated with at least 2 prior systemic therapies for FL
* Radiographically measurable lymphadenopathy or extranodal lymphoid malignancy (defined as the presence of ≥ 1 lesion that measures > 1.5 cm in the LD and ≥ 1.0 cm in the LPD, respectively) as assessed by CT or MRI
* Participants must be willing to undergo an incisional, excisional, or core needle lymph node or tissue biopsy or provide a lymph node or tissue biopsy collected after the completion of last therapy. An earlier archived lymph node or tissue biopsy is acceptable if hospitalization is required for biopsy (eg. no superficial lymph node) and SUVmax by FDG-PET is < 14
* ECOG performance status 0 to 2
* Life expectancy ≥ 12 weeks
* Adequate hematologic, hepatic, and renal functions ANC ≥ 1.0 × 109/L Hemoglobin ≥ 8.0 g/dL. Platelet count ≥ 50 × 109/L. Total bilirubin ≤ 1.5 × ULN. Participants with documented history of Gilbert's syndrome and in whom total bilirubin elevations are accompanied by elevated indirect bilirubin are eligible.

ALT/AST ≤ 2.5× ULN or ≤ 5 × ULN in the presence of liver involvement. Calculated creatinine clearance ≥ 40 mL/min by the Cockcroft-Gault Equation or the estimated glomerular filtration rate ≥ 40 mL/min/1.73 m2 using the Modification of Diet in Renal Disease formula.

* Female participants agree to use medically acceptable contraceptive measures, should not be breastfeeding, and must have a negative pregnancy test before the start of study drug administration.
* Female participants of childbearing potential must understand and accept that pregnancy must be avoided during participation in the study.
* Male participants should avoid fathering children from screening through at least 93 days after the last dose of study treatment.

Exclusion Criteria:

* Known histological transformation from indolent NHL to DLBCL
* History of central nervous system lymphoma (either primary or metastatic)
* Prior treatment with the following:

  1. Selective PI3Kδ or pan-PI3K inhibitors (eg, idelalisib, copanlisib, duvelisib, etc).
  2. Bruton's tyrosine kinase inhibitor (eg, ibrutinib).
* Allogeneic SCT within the last 6 months, or autologous SCT within the last 3 months before the date of study treatment administration
* Active graft-versus-host disease
* Use of immunosuppressive therapy within 28 days of the date of study treatment administration
* Concurrent anticancer therapy
* Significant concurrent, uncontrolled medical condition including, but not limited to, renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, neurological, cerebral, or psychiatric disease
* Current or previous other malignancy within 3 years of study entry, except cured basal or squamous cell skin cancer, superficial bladder cancer, prostate intraepithelial neoplasm, carcinoma in situ of the cervix, or other noninvasive or indolent malignancy without sponsor approval.
* Hepatitis B (HBV) or HCV infection
* Current New York Heart Association Class II to IV congestive heart failure or uncontrolled arrhythmia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2023-02-16 (Actual); Study Completion 2023-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Incyte Medical Monitor, Study Director — Incyte Biosciences Japan GK
Locations (30):
- Japan (30):
  - Ja-Aichi Anjo Kosei Hospital, Anjo
  - University of Fukui Hospital, Fukui
  - Jcho Kyushu Hospital, Fukuoka
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Fukushima Medical University Hospital, Fukushima
  - Kansai Medical University Hospital, Hirakata
  - Hokuyukai Sapporo Hokuyu Hospital, Hokkaido
  - Hyogo College of Medicine Hospital, Hyōgo
  - Nho Mito Medical Center, Ibaraki
  - Tokai University Hospital, Isehara
  - Jiaikai Imamura General Hospital, Kagoshima
  - Kobe City Medical Center General Hospital, Kobe
  - University Hospital Kyoto Prefectural University of Medicine, Kyoto
  - Nho Matsumoto Medical Center, Matsumoto
  - Nho Shikoku Cancer Center, Matsuyama
  - Nagano Red Cross Hospital, Nagano
  - National Hospital Organization Nagoya Medical Center, Nagoya
  - Japanese Red Cross Nagoya Daini Hospital, Nagoya
  - Red Cross Nagoya Daini Hospital, Nagoya
  - Tenri Hospital, Nara
  - Miyagi Cancer Center, Natori
  - Niigata Cancer Center Hospital, Niigata
  - Okayama University Hospital, Okayama
  - Ogaki Municipal Hospital, Ōgaki
  - Nho Hokkaido Cancer Center, Sapporo
  - Tohoku University Hospital, Sendai
  - Shizuoka Cancer Center, Shizuoka
  - Nippon Medical School Hospital, Tokyo
  - Yokohama Municipal Citizens Hospital, Yokohama
  - Yokohama City University Medical Center, Yokohama

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

REFERENCES:
- [Derived] Fukuhara N, Yoshida I, Ishiguro T, Fujimoto K, Kuroda J, Uchida T, Yamamoto R, Ogawa Y, Hiramatsu Y, Ito T, Katagiri S, Nakazato T, Suzukawa K, Kinami K, Zhou M, Negoro E. PI3Kdelta Inhibitor Parsaclisib in Japanese Patients With Relapsed or Refractory Follicular Lymphoma. Cancer Sci. 2025 Aug;116(8):2189-2197. doi: 10.1111/cas.70046. Epub 2025 May 14. PMID 40365847

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was conducted at 19 study centers in Japan.
Groups:
- Parsaclisib 20 mg/2.5 mg: Participants received parsaclisib 20 milligrams (mg) once daily for 8 weeks, followed by 2.5 mg once daily, continuously. Participants received treatment until disease progression, death, hematopoietic stem cell transplantation (HSCT) (if eligible), unacceptable toxicity, or consent withdrawal.
Period: Overall Study
Arm/Group | Parsaclisib 20 mg/2.5 mg
Started | 42
Completed | 0
Not Completed | 42
Not completed — Death | 4
Not completed — Withdrawal by Subject | 1
Not completed — Transitioned to Rollover Study | 19
Not completed — Progressive Disease | 18

BASELINE CHARACTERISTICS:
Arm/Group | Parsaclisib 20 mg/2.5 mg
Number analyzed (Participants) | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.5 (7.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 42
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Target lesion size, as determined by Independent Review Committee and the Investigator [Mean (Standard Deviation); unit: millimeters squared (mm^2)] — Target lesion size was measured by the sum of the products of the diameters of all target lesion sizes. Population: Only participants with available data (who had measurable regions) were analyzed.
  millimeters squared (mm^2)
    Independent Review Committee: number analyzed (Participants) | 41
    Independent Review Committee | 2210.12 (1456.044)
    Investigator | 2487.24 (2197.143)

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants with a complete response (CR) or partial response (PR) as defined by revised response criteria for lymphoma, as determined by an Independent Review Committee (IRC). CR: target nodes/nodal masses regressed to ≤1.5 centimeters (cm) in the longest transverse diameter (LDi); no nonmeasured lesions; regression to normal for organ enlargement; no new lesions; and normal bone marrow by morphology and negative immunohistochemistry if indeterminate. PR: ≥50% decrease in sum of the product of the diameters (SPD) of up to 6 target measurable nodes and extranodal sites; absent/regressed nonmeasured lesions (but no increase); spleen regressed by >50% in length beyond normal; and no new lesions.
Time Frame: up to approximately 3 years
Population: Full Analysis Set: all participants enrolled in the study who received at least 1 dose of parsaclisib. Confidence intervals were calculated based on the exact method for binomial distributions.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Parsaclisib 20 mg/2.5 mg
Number analyzed (Participants) | 42
percentage of participants | 88.1 [74.4 to 96.0]

2. Secondary Outcome: Complete Response Rate (CRR)
Description: CRR was defined as the percentage of participants with a CR as defined by revised response criteria for lymphoma, as determined by an IRC. CR was defined as: target nodes/nodal masses regressed to ≤1.5 cm in the LDi; no nonmeasured lesions; regression to normal for organ enlargement; no new lesions; and normal bone marrow by morphology and negative immunohistochemistry if indeterminate.
Time Frame: up to approximately 3 years
Population: Full Analysis Set. Confidence intervals were calculated based on the exact method for binomial distributions.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Parsaclisib 20 mg/2.5 mg
Number analyzed (Participants) | 42
percentage of participants | 23.8 [12.1 to 39.5]

3. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the time from the first documented evidence of CR or PR until disease progression or death from any cause among participants who achieved an objective response, as determined by radiographic disease assessment provided by an IRC. Progressive disease was defined as ≥1 of the following: abnormal individual node/lesion meeting specific criteria; new/recurrent splenomegaly; new/clear progression of pre-existing nonmeasured lesions; regrowth of any previously resolved lesions; new node >1.5 cm in any axis; new extranodal site >1.0 cm in any axis; assessable disease of any size attributable to lymphoma; new/recurrent involvement of bone marrow.
Time Frame: up to 20.0 months
Population: Full Analysis Set. Only participants with a CR or PR were analyzed. The 95% confidence interval was calculated using the generalization of Brookmeyer and Crowley's method with log-log transformation.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Parsaclisib 20 mg/2.5 mg
Number analyzed (Participants) | 37
months | NA [8.02 to NA] — The median and the upper limit of the confidence interval were not estimable because too few participants had disease progression or died.

4. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time from the date of the first dose of study treatment until the earliest date of disease progression, as determined by radiographic disease assessment provided by an IRC, or death from any cause. Progressive disease was defined as any new lesion or increase by ≥ 50% of previously involved sites from nadir.
Time Frame: up to approximately 3 years
Population: Fully Analysis Set. The 95% confidence interval was calculated using the generalization of Brookmeyer and Crowley's method with log-log transformation.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Parsaclisib 20 mg/2.5 mg
Number analyzed (Participants) | 42
months | NA [11.17 to NA] — The median and the upper limit of the confidence interval were not estimable because too few participants had disease progression or died.

5. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from the date of the first dose of study treatment until death from any cause.
Time Frame: up to approximately 3 years
Population: Full Analysis Set. The 95% confidence interval was calculated using the generalization of Brookmeyer and Crowley's method with log-log transformation.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Parsaclisib 20 mg/2.5 mg
Number analyzed (Participants) | 42
months | NA [23.06 to NA] — The median and the upper limit of the confidence interval were not estimable because too few participants died.

6. Secondary Outcome: Best Percentage Change in Target Lesion Size From Baseline, as Determined by Independent Review Committee and the Investigator
Description: Target lesion size was measured by the sum of the products of the diameters of all target lesion sizes. The best percent change from Baseline was defined as the largest decrease, or smallest increase if no decrease, from Baseline in target lesion sizes on/before new anti-lymphoma therapy during the study. Percentage change was calculated as ([the post-Baseline value minus the Baseline value] / the Baseline value) x 100.
Time Frame: up to approximately 3 years
Population: Full Analysis Set. Only participants with available data (who had measurable regions) were analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Parsaclisib 20 mg/2.5 mg
Number analyzed (Participants) | 42
percent change
  Independent Review Committee: number analyzed (Participants) | 41
  Independent Review Committee | -67.26 (39.897)
  Investigator | -79.31 (23.181)

7. Secondary Outcome: Number of Participants With Any Treatment-emergent Adverse Event (TEAE)
Description: An adverse event was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug-related. An AE could therefore have been any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study treatment. A TEAE was defined as any AE either reported for the first time or the worsening of a pre-existing event after the first dose of study drug and within 30 days of the last administration of study drug.
Time Frame: up to 1041 days
Population: Safety Population: all enrolled participants who received at least 1 dose of parsaclisib
Measure: Count of Participants; unit: Participants
Arm/Group | Parsaclisib 20 mg/2.5 mg
Number analyzed (Participants) | 42
Participants | 42

8. Secondary Outcome: Number of Participants With Any Grade 3 or Higher TEAE
Description: An adverse event was as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug-related. A TEAE was defined as any AE either reported for the first time or the worsening of a pre-existing event after the first dose of study drug and within 30 days of the last administration of study drug. The severity of AEs was assessed using Common Terminology Criteria for Adverse Events (CTCAE) v5.0. Grade 1: mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; treatment not indicated. Grade 2: moderate; minimal, local, or noninvasive treatment indicated; limiting age appropriate activities of daily living. Grade 3: severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care activities of daily living. Grade 4: life-threatening consequences; urgent treatment indicated. Grade 5: fatal.
Time Frame: up to 1041 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Parsaclisib 20 mg/2.5 mg
Number analyzed (Participants) | 42
Participants | 28

ADVERSE EVENTS:
Time Frame: up to 1041 days
Description: Treatment-emergent adverse events (TEAE ), defined as any adverse events either reported for the first time or the worsening of pre-existing events after the first dose of study drug and within 30 days of the last administration of study drug, have been reported.
Groups:
- Total: Total
Arm/Group | Parsaclisib 20 mg/2.5 mg | Total
All-Cause Mortality (participants affected / at risk) | 4/42 | 4/42
Serious Adverse Events (participants affected / at risk) | 15/42 | 15/42
Other Adverse Events (participants affected / at risk) | 38/42 | 38/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Parsaclisib 20 mg/2.5 mg (N=42) | Total (N=42)
Aortic aneurysm (Vascular disorders) | 1 (1) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
COVID-19 (Infections and infestations) | 2 (3) | 2 (3)
Cardiac failure (Cardiac disorders) | 2 (2) | 2 (2)
Cataract (Eye disorders) | 1 (2) | 1 (2)
Cheilitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Cytomegalovirus colitis (Infections and infestations) | 2 (2) | 2 (2)
Cytomegalovirus enteritis (Infections and infestations) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 1 (1)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 3 (3) | 3 (3)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Urethritis (Infections and infestations) | 1 (1) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Parsaclisib 20 mg/2.5 mg (N=42) | Total (N=42)
Alanine aminotransferase increased (Investigations) | 4 (6) | 4 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 5 (5)
Aspartate aminotransferase increased (Investigations) | 4 (6) | 4 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4)
Conjunctivitis (Infections and infestations) | 3 (3) | 3 (3)
Constipation (Gastrointestinal disorders) | 8 (8) | 8 (8)
Cytomegalovirus infection reactivation (Infections and infestations) | 6 (6) | 6 (6)
Decreased appetite (Metabolism and nutrition disorders) | 4 (5) | 4 (5)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 11 (21) | 11 (21)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3)
Eczema (Skin and subcutaneous tissue disorders) | 5 (6) | 5 (6)
Herpes zoster (Infections and infestations) | 5 (5) | 5 (5)
Hypertension (Vascular disorders) | 4 (4) | 4 (4)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 (3) | 3 (3)
Hypogammaglobulinaemia (Immune system disorders) | 3 (3) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (4) | 4 (4)
Nausea (Gastrointestinal disorders) | 4 (5) | 4 (5)
Neutropenia (Blood and lymphatic system disorders) | 5 (12) | 5 (12)
Neutrophil count decreased (Investigations) | 9 (28) | 9 (28)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5) | 5 (5)
Stomatitis (Gastrointestinal disorders) | 8 (11) | 8 (11)
Oedema peripheral (General disorders) | 3 (3) | 3 (3)
Pyrexia (General disorders) | 3 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (2):
  • Study Protocol (2023-01-24): https://cdn.clinicaltrials.gov/large-docs/37/NCT04434937/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-26): https://cdn.clinicaltrials.gov/large-docs/37/NCT04434937/SAP_001.pdf